CLINICAL TRIAL: NCT07000071
Title: Non-invasive Secondary Respiratory Support in Late Preterm and Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Assistant professor of Pediatrics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201275
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-01

CONDITIONS: Neonates; Respiratory Distress; Non- Invasive Ventilation
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nasal Continuous positive airway pressure (NCPAP) (Active Comparator): apply continuous positive airway pressure using nasopharyngeal interface. positive end expiratory pressure (PEEP ) used 5-7 cm H2O. Neonates will be supported with NCPAP following extubation.
  Interventions: Device: NCPAP
- Nasal intermittent pressure ventilation (NIPPV) (Active Comparator): Neonates will be supported with NIPPV following extubation.
  Interventions: Device: NIPPV
- Nasal high frequency ventilation (NHFOV) (Active Comparator): Neonates will be supported with NHFOV following extubation. stating mean airway pressure 8 and can reach upto 15 cm H2O Delta pressure used is 20 Frequency 10 HZ
  Interventions: Device: NHFOV

INTERVENTIONS:
Device: NCPAP — Apply nasal continuous positive airway pressure in intubated patients with respiratory distress at time of weaning
  Arms: Nasal Continuous positive airway pressure (NCPAP)
Device: NIPPV — Apply nasal intermittent positive pressure ventilation in intubated patients with respiratory distress at time of weaning
  Arms: Nasal intermittent pressure ventilation (NIPPV)
Device: NHFOV — Apply nasal high frequency ventilation in intubated patients with respiratory distress at time of weaning
  Arms: Nasal high frequency ventilation (NHFOV)

SUMMARY:
The aim of the present work is to compare between various modes of non-invasive respiratory support (including NCPAP, NIPPV, and NHFOV) as secondary respiratory support modes in late preterm and term neonates as regards the need for reintubation. Additionally, the study aims at comparing between the three modes concerning the associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age (GA) is between 34 and 41 weeks.
* Extubation from invasive mechanical ventilation initiated due to RD, irrespective to the cause of RD.
* Respiratory distress is assessed based on clinical manifestations (tachypnea, nasal flaring, intercostal retractions, diminished air entry, and or grunting)

Exclusion Criteria:

* Major congenital anomalies.
* Major cardiac diseases.
* Presence of cardiovascular instability (sepsis, severe dehydration, severe anemia).
* Neurologically insulted neonates who are unable to take adequate spontaneous breathing.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Failure rate | 72 hours after weaning
  need for reintubation and invasive mechanical ventilation

SECONDARY OUTCOMES:
duration of non-invasive ventilation | first 72 hours after weaning from mechanical ventillation
  duration of noninvasive ventilation till patients become weaned to free flow oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Mohamed Farag, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided